CLINICAL TRIAL: NCT00221221
Title: Physical Activity Promotion in Breast Cancer Survivors: A Population Based Randomized Controlled Trial
Brief Title: Physical Activity Promotion in Breast Cancer Survivors
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: ACTION
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: breast cancer survivors; physical activity; health promotion
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

INTERVENTIONS:
Device: Pedometer
Device: Exercise guidebook

SUMMARY:
Over 30 studies have shown that exercise can improve physical fitness, reduce fatigue, increase functioning, and enhance overall quality of life (QoL) in breast cancer survivors both during and after treatments. Research has also shown, however, that breast cancer survivors experience a significant reduction in physical activity during treatments that is not recovered even years after treatments are completed. The objectives of this study are to examine the effects of two behavior change interventions (a step pedometer and printed materials) on physical activity, social cognitive variables, and QoL in a population-based sample of breast cancer survivors. Approximately 300 breast cancer survivors living in Northern Alberta will be randomized to one of four groups: (1) an exercise recommendation only group (viewed as the current standard of care), (2) an exercise recommendation plus pedometer group, (3) an exercise recommendation plus printed materials group, and (4) an exercise recommendation plus pedometer and printed materials group. Our primary hypothesis is that participants receiving the combined pedometer and printed materials intervention will report the greatest change in physical activity. Our secondary hypotheses are that these interventions will also result in improved QoL and more positive social cognitive beliefs about exercise in breast cancer survivors. Given the geographic dispersion of our population, finding practical and sustainable interventions that employ distance medicine-based approaches may be ideal for promoting healthy activity patterns in breast cancer survivors in Northern Alberta.

DETAILED DESCRIPTION:
Approximately 300 breast cancer survivors living in Northern Alberta will be randomized to one of four groups: (1) an exercise recommendation only group (viewed as the current standard of care), (2) an exercise recommendation plus pedometer group, (3) an exercise recommendation plus printed materials group, and (4) an exercise recommendation plus pedometer and printed materials group. Our primary hypothesis is that participants in the three intervention groups will report a greater positive change in physical activity than participants in the exercise recommendation only group. Furthermore, we expect that participants receiving the combined pedometer and printed materials intervention will report the greatest change in physical activity. Our secondary hypotheses are that these interventions will also result in improved QoL and more positive social cognitive beliefs about exercise in breast cancer survivors. Our sample size was determined by a power calculation. Based on the literature, we believe that an increase of 2,000 steps per day is a meaningful change that will result in health benefits for breast cancer survivors. We estimate a standard deviation of about 4,000 steps per day. Therefore, to detect a medium standardized effect (d = .50) with a power of .80 and a two-tailed alpha <.05, we need 63 participants per group. To account for a possible 15% loss to follow up, we will randomize 75 participants to each group. Our printed materials will be developed based on the tenets of the theory of planned behavior and will include activities designed to enhance instrumental and affective attitudes, injunctive and descriptive norms, and self-efficacy and perceptions of control. These materials will be developed based on our previous research identifying the key beliefs that should be targeted in a theory of planned behavior-based intervention.

Our procedure will be to identify and screen potential participants for eligibility through the Alberta Cancer Registry. After obtaining written informed consent from the individual's treating oncologist, all eligible participants will be sent a letter of invitation to participate in the study. Interested participants will complete a baseline questionnaire that will include measures of physical activity (the Godin Leisure-Time Exercise Questionnaire), QoL (Functional Assessment of Cancer Therapy-Breast and Anemia), and social cognitive variables from the theory of planned behavior (based on the guidelines from Ajzen and our previous research). Participants will also wear a pedometer for a 7-day monitoring period to obtain baseline steps. Participants will then be randomized to one of four groups. Depending on randomization, the participants will then receive the appropriate materials. All groups will be recommended to accumulate at least 30 minutes of moderate intensity physical activity at least five days per week which would result in about 15,000 steps per week (or 2,000 steps per day). At the end of the 12-week intervention period, all participants will complete the same post intervention questionnaire and undergo another 7-day monitoring period to obtain step values. Participants will be contacted at 6 months for follow-up and complete the same questionnaire for a final time.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed breast cancer.
* mentally competent.
* physician approval to participate in the study.
* free from chronic medical and orthopaedic conditions.
* no current or planned pregnancy.
* ability to read and understand English.
* must be in the post treatment phase of their cancer trajectory.
* willing to accept random assignment.
* not currently participating in another QoL intervention.
* no known or active metastatic disease.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2005-07; Study Completion 2006-03

PRIMARY OUTCOMES:
Exercise behavior

SECONDARY OUTCOMES:
Quality of life
Social cognitive determinants of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey KH Vallance, MA, Principal Investigator — University of Alberta; Kerry S Courneya, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Behavioral Medicine Laboratory, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Vallance JK, Courneya KS, Plotnikoff RC, Yasui Y, Mackey JR. Randomized controlled trial of the effects of print materials and step pedometers on physical activity and quality of life in breast cancer survivors. J Clin Oncol. 2007 Jun 10;25(17):2352-9. doi: 10.1200/JCO.2006.07.9988. PMID 17557948